CLINICAL TRIAL: NCT03199846
Title: Treatment Patterns and Outcomes Study in Patients With Unresectable Stage III and Metastatic (Stage IV) Melanoma in the United States
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-983
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- advanced melanoma patients: Part 1 will consist of a representative sample of advanced melanoma patients, irrespective of date of diagnosis of stage III unresectable and metastatic/stage IV, to address information objectives on treatment patterns, clinical outcomes, and resource use after the start of treatment post-launch of new drugs, ie, since 2011 for ipi and 2015 for ipi + nivo in advanced melanoma
  Interventions: Other: Non-Interventional
- Ipi monotherapy: Part 2: patients must have been prescribed Ipi monotherapy during the index period between 01-Jan-2015 and 31-May-2016.
  Interventions: Other: Non-Interventional
- Ipi + nivo combination therapy: Part 2: patients must have been prescribed Ipi + nivo combination therapy during the index period between 01-Jan-2015 and 31-May-2016.
  Interventions: Other: Non-Interventional
- Dabrafenib + trametinib combination therapy: Part 2: patients must have been prescribed Dabrafenib + trametinib combination therapy during the index period between 01-Jan-2015 and 31-May-2016.
  Interventions: Other: Non-Interventional
- Pembro monotherapy: Part 2: patients must have been prescribed Pembro monotherapy during the index period between 01-Jan-2015 and 31-May-2016
  Interventions: Other: Non-Interventional
- Nivo monotherapy: Part 2: patients must have been prescribed Nivo monotherapy during the index period between 01-Jan-2015 and 31-May-2016
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study will collect real-world data from advanced melanoma diagnosis through most recent visit and data sourced from patient medical records following a 2-part study design consisting of a random sample (Part 1) and an oversample (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Diagnosis of unresectable stage III and/or metastatic (stage IV) melanoma before 01-Nov-2015
* Initiating a new line of therapy during the index period between 01-Jan-2015 and 31-May-2016, irrespective of advanced melanoma diagnosis date
* Medical history available for medical chart abstraction from date of diagnosis through most recent or current therapy (defined as end of data collection period)

Exclusion Criteria:

* Physicians unwilling or unable to follow study instructions
* Patients who were previously enrolled in a cancer treatment-related clinical trial since the diagnosis of unresectable stage III and/or metastatic (stage IV) melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initiating a new line of therapy for unresectable stage III and/or metastatic (stage IV) melanoma during the index period between 01-Jan-2015 and 31-May-2016.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Distribution of treatment patterns for advanced melanoma patients | Aproximately 6 months
  Distribution of treatment patterns for advanced melanoma patients including, treatment regimen selection and rationale, as well as time to initiation of therapy and type of therapy

SECONDARY OUTCOMES:
Distribution of prescribing patterns | Approximately 16 months
  Distribution of prescribing patterns by type of practice setting and melanoma patient volume
Distribution of Patient Age at index date | at baseline
  Patient Age at index date will be determined from Medical Records
Distribution of Patient's Sex at Index Date | At Baseline
  Patient's sex will be determined from Medical Records
Distribution of Comorbidities at index date | At Baseline
  Comorbidities will be determined using the Charlson Comorbidity Index (CCI)
Distribution of Healthcare Coverage type | At Baseline
  Healthcare Coverage type will be determined using Medical Records
Distribution of Diagnosis Date | At Baseline
  Melanoma Diagnosis Date will be determined using medical records
Distribution of Advanced Diagnosis Date | At Baseline
  Date of advanced/ metastatic melanoma diagnosis will be determined using medical records
Distribution of Age at Onset | At Baseline
  Diagnosis date-Date of Birth
Distribution of Disease stage at time of diagnosis | At Baseline
  Disease stage at time of diagnosis will be determined using medical records
Distribution of Disease stage at subsequent visits | Approximately 16 months
  Disease stage at subsequent visits will be determined using medical records
Distribution of ECOG status at Baseline | At Baseline
  Eastern Cooperative Oncology Group (ECOG) status at Baseline will be determined using medical records
Distribution of ECOG status at Last Visit | Approximately 16 months
  Eastern Cooperative Oncology Group (ECOG) status at Last Visit will be determined using medical records
Distribution of Biomarker status at baseline | at baseline
  Biomarker status will be determined using Medical Records
Distribution of treatment-related adverse events | Approximately 16 months
  treatment-related adverse events will be determined using medical records
Distribution of Overall Survival (OS) from Advanced Diagnosis | Approximately 16 months
  Date of death minus advanced/metastatic diagnosis date, censoring for LTF or end of observation
Distribution of Progression-Free Survival (PFS) at Advanced Diagnosis | Approximately 16 months
  Date of progression (increase in tumor size or increase in cancer stage)/start of next line of therapy minus advanced/metastatic diagnosis date, censoring for LTF or end of observation
Distribution of Overall Response Rate (ORR) | Approximately 16 months
Distribution of Overall Survival (OS) from Index Date | Approximately 16 months
  Date of death minus index treatment start date, censoring for LTF or end of observation
Distribution of Progression-Free Survival (PFS) at Index Date | Approximately 16 months
  Date of progression (increase in tumor size or increase in cancer stage)/start of next line of therapy minus index treatment start date, censoring for LTF or end of observation
Distribution of melanoma related HCRU | Approximately 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Morristown, New Jersey, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx